CLINICAL TRIAL: NCT01861301
Title: A Phase 2 Study of ARQ 197 in Patients With Previously-Treated Malignant Mesothelioma
Brief Title: Tivantinib in Treating Patients With Previously Treated Malignant Mesothelioma
Status: Terminated | Phase: Phase 2 | Type: Interventional
Sponsor: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: NCI-2013-00937; NCI-2013-00937 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); 12-2158; 12-2158 (Other: University of Chicago Comprehensive Cancer Center); 9267 (Other: CTEP); N01CM00071 (NIH); P30CA014599 (NIH)
Record Dates: First submitted 2013-05-20; First posted 2013-05-23 (Estimated); Results first posted 2016-10-24 (Estimated); Last update posted 2016-10-24 (Estimated); Status verified 2016-08

CONDITIONS: Epithelioid Mesothelioma; Recurrent Malignant Mesothelioma; Sarcomatoid Mesothelioma; Stage II Pleural Mesothelioma; Stage III Pleural Mesothelioma; Stage IV Pleural Mesothelioma
MeSH Terms: conditions — Mesothelioma, Malignant; Solitary Fibrous Tumor, Pleural | interventions — ARQ 197

ARMS (1):
- Treatment (tivantinib) (Experimental): Patients receive tivantinib 360 PO BID. Treatment continues in the absence of disease progression or unacceptable toxicity.
  Interventions: Other: Laboratory Biomarker Analysis; Drug: Tivantinib

INTERVENTIONS:
Other: Laboratory Biomarker Analysis — Correlative studies
Drug: Tivantinib — Given PO
  Other Names: ARQ 197; ARQ-197; c-Met Inhibitor ARQ 197

SUMMARY:
This phase II trial studies how well tivantinib works in treating patients with previously treated malignant mesothelioma. Tivantinib may stop the growth of tumor cells by blocking some of the enzymes needed for cell growth.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. To determine the objective response rate of patients with malignant mesothelioma who are treated with ARQ 197 (tivantinib).

SECONDARY OBJECTIVES:

I. To determine the progression-free survival of patients with malignant mesothelioma who are treated with ARQ 197.

II. To determine the toxicity experienced by patients with malignant mesothelioma who are treated with ARQ 197.

III. To determine median and overall survival of patients with malignant mesothelioma who are treated with ARQ 197.

TERTIARY OBJECTIVES:

I. To determine the frequency of mesenchymal-epithelial transition (MET) gene amplification in malignant mesothelioma patient tumor samples, and to correlate the results with MET immunohistochemistry (IHC).

II. To determine whether MET gene amplification results in increased sensitivity to ARQ 197 as observed by improved clinical outcomes (response rate [RR] and progression free survival [PFS]) compared to those without MET gene over-expression/amplification.

III. To determine whether high baseline serum hepatocyte growth factor (HGF), as well as changes in serum HGF during treatment at pre-defined early time points, correlate with treatment efficacy and clinical outcome, as measured by response rate and progression-free survival.

IV. To identify mutations by sequencing of specific areas of the MET gene in tumor samples (semaphorin [SEMA], jumonji [JM] and tyrosine kinase domains).

V. To perform immunohistochemistry (IHC) of mesothelioma tumors for HGF, MET and phosphorylated (p)-MET (pY1003 and pY1230/34/35).

VI. To assess serum HGF and serum soluble MET levels by enzyme linked immunosorbent assay (ELISA) (R&D systems) pre-treatment, after 2 cycles and at disease progression.

OUTLINE:

Patients receive tivantinib orally (PO) twice daily (BID). Treatment continues in the absence of disease progression or unacceptable toxicity.

After completion of study treatment, patients are followed up for 1 year.

ELIGIBILITY:
Inclusion Criteria:

* Patients must have histologically or cytologically confirmed malignant pleural or peritoneal mesothelioma, epithelial, sarcomatoid, or mixed subtype; the patient's disease must be metastatic, recurrent, or unresectable
* Patients must have measurable disease, defined as at least one lesion that can be accurately measured in at least one dimension (longest diameter to be recorded for non-nodal lesions and short axis for nodal lesions) as >= 20 mm with conventional techniques or as >= 10 mm with spiral computed tomography (CT) scan, magnetic resonance imaging (MRI), or calipers by clinical exam; pleural effusions and ascites are not considered measurable lesions
* No more than two prior cytotoxic chemotherapy regimens; prior chemotherapy with pemetrexed is required; prior intrapleural cytotoxic agents (including bleomycin) are allowed, and are not counted as a cytotoxic chemotherapy; chemotherapy must have been completed at least 4 weeks prior; patients who have previously received radiation therapy are eligible provided that the only site of measurable disease is not located within the radiation therapy port; at least 4 weeks must have elapsed from completion of the radiation therapy and all signs of toxicity must have resolved
* Eastern Cooperative Oncology Group (ECOG) performance status =< 1 (Karnofsky >= 70%)
* Life expectancy of greater than 3 months
* Hemoglobin >= 9.0 g/dL
* White blood cells (WBC) >= 3,000/mcL
* Absolute neutrophil count >= 1,500/mcL
* Platelets >= 100,000/mcL
* Total bilirubin =< 1.5 X institutional upper limit of normal
* Aspartate aminotransferase (AST) (serum glutamic oxaloacetic transaminase [SGOT])/alanine aminotransferase (ALT) (serum glutamate pyruvate transaminase [SGPT]) =< 2.5 X institutional upper limit of normal
* Serum creatinine =< 1.5 X institutional upper limit of normal OR creatinine clearance >= 60 mL/min/1.73 m^2 for patients with creatinine levels above institutional normal
* The effects of ARQ 197 on the developing human fetus are unknown; for this reason and because tyrosine kinase inhibitors as well as other therapeutic agents used in this trial are known to be teratogenic, women of child-bearing potential and men must agree to use adequate contraception (hormonal or barrier method of birth control; abstinence) prior to study entry and for the duration of study participation; should a woman become pregnant or suspect she is pregnant while she or her partner is participating in this study, she should inform her treating physician immediately; men treated or enrolled on this protocol must also agree to use adequate contraception prior to the study, for the duration of study participation, and 4 months after completion of ARQ 197 administration
* Ability to understand and the willingness to sign a written informed consent document

Exclusion Criteria:

* Patients who have had chemotherapy or radiotherapy within 4 weeks (6 weeks for nitrosoureas or mitomycin C) prior to entering the study or those who have not recovered from adverse events (to grade =< 1) due to agents administered more than 4 weeks earlier
* Patients who are receiving any other investigational agents
* Patients with known brain metastases should be excluded from this clinical trial because of their poor prognosis and because they often develop progressive neurologic dysfunction that would confound the evaluation of neurologic and other adverse events
* History of allergic reactions attributed to compounds of similar chemical or biologic composition to ARQ 197
* ARQ 197 is metabolized by cytochrome P450 (CYP)2C19, and to a lesser extent CYP3A4; the metabolism and consequently overall pharmacokinetics of ARQ 197 could be altered by inhibitors and/or inducers or other substrates of CYP2C19 and CYP3A4; while inhibitors/inducers of these cytochrome P450 isoenzymes are not specifically excluded, investigators should be aware that ARQ 197 exposure may be altered by the concomitant administration of these drugs; because the lists of these agents are constantly changing, it is important to regularly consult a frequently-updated list; as part of the enrollment/informed consent procedures, the patient will be counseled on the risk of interactions with other agents, and what to do if new medications need to be prescribed or if the patient is considering a new over-the-counter medicine or herbal product
* History of congestive heart failure defined as Class II to IV per New York Heart Association (NYHA) classification; active coronary artery disease (CAD); clinically significant bradycardia or other uncontrolled, cardiac arrhythmia defined as >= grade 3 according to National Cancer Institute (NCI) Common Terminology Criteria for Adverse Events (CTCAE), version 4.0, or uncontrolled hypertension; myocardial infarction occurring within 6 months prior to study entry (myocardial infarction occurring > 6 months prior to study entry is permitted)
* Uncontrolled intercurrent illness including, but not limited to, ongoing or active infection, symptomatic congestive heart failure, unstable angina pectoris, cardiac arrhythmia, or psychiatric illness/social situations that would limit compliance with study requirements
* Pregnant women are excluded from this study because ARQ 197 is a tyrosine kinase inhibitor with the potential for teratogenic or abortifacient effects; because there is an unknown but potential risk for adverse events in nursing infants secondary to treatment of the mother with ARQ 197, breastfeeding should be discontinued if the mother is treated with ARQ 197
* Human immunodeficiency virus (HIV)-positive patients on combination antiretroviral therapy are ineligible because of the potential for pharmacokinetic interactions with ARQ197; in addition, these patients are at increased risk of lethal infections when treated with marrow-suppressive therapy; appropriate studies will be undertaken in patients receiving combination antiretroviral therapy when indicated
* No prior treatment with a c-MET inhibitor

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 18 (Actual)
Dates: Start 2013-01; Primary Completion 2015-03 (Actual); Study Completion 2015-03 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Hedy Kindler, Principal Investigator — University of Chicago Comprehensive Cancer Center
Locations (18):
- United States (18):
  - City of Hope Comprehensive Cancer Center, Duarte, California
  - USC / Norris Comprehensive Cancer Center, Los Angeles, California
  - University of California Davis Comprehensive Cancer Center, Sacramento, California
  - City of Hope South Pasadena, South Pasadena, California
  - Northwestern University, Chicago, Illinois
  - University of Chicago Comprehensive Cancer Center, Chicago, Illinois
  - Decatur Memorial Hospital, Decatur, Illinois
  - NorthShore University HealthSystem-Evanston Hospital, Evanston, Illinois
  - Ingalls Memorial Hospital, Harvey, Illinois
  - Illinois CancerCare-Peoria, Peoria, Illinois
  - Southern Illinois University School of Medicine, Springfield, Illinois
  - Fort Wayne Medical Oncology and Hematology Inc-Parkview, Fort Wayne, Indiana
  - Indiana University/Melvin and Bren Simon Cancer Center, Indianapolis, Indiana
  - University of Michigan Comprehensive Cancer Center, Ann Arbor, Michigan
  - Wayne State University/Karmanos Cancer Institute, Detroit, Michigan
  - Mercy Hospital Saint Louis, St Louis, Missouri
  - Penn State Milton S Hershey Medical Center, Hershey, Pennsylvania
  - University of Pittsburgh Cancer Institute, Pittsburgh, Pennsylvania

RESULTS

PARTICIPANT FLOW:
Groups:
- Treatment (Tivantinib): Patients receive tivantinib 360 mg PO BID. Treatment continues in the absence of disease progression or unacceptable toxicity.
Period: Overall Study
Arm/Group | Treatment (Tivantinib)
Started | 18
Completed | 18
Not Completed | 0

BASELINE CHARACTERISTICS:
Arm/Group | Treatment (Tivantinib)
Number analyzed (Participants) | 18
Age, Continuous [Median (Full Range); unit: years] | 66.5 [19 to 81]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 7
  Male | 11
Region of Enrollment [Number; unit: participants]
  United States | 18

OUTCOME MEASURES:

1. Primary Outcome: Objective Radiologic Response Rate (Complete or Partial Response) Assessed by the Response Evaluation Criteria in Solid Tumors (RECIST) v1.1
Description: Per Response Evaluation Criteria In Solid Tumors Criteria (RECIST v1.1) for target lesions and assessed by CT or MRI: Complete Response (CR), Disappearance of all target lesions; Partial Response (PR), >=30% decrease in the sum of the longest diameter of target lesions; Overall Response (OR) = CR + PR.
Time Frame: Up to 1 year
Population: Note: Study terminated for futility due to insufficient number of objective responders in first stage.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Treatment (Tivantinib)
Number analyzed (Participants) | 18
percentage of participants | 0 [0 to 18.5]

2. Secondary Outcome: Incidence of Adverse Events, Graded Per NCI CTCAE Version 4
Description: Grade 3 or higher AE of any type, regardless of attribution.
Time Frame: Up to 2 years
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Treatment (Tivantinib)
Number analyzed (Participants) | 18
percentage of participants | 22.2 [6.4 to 47.6]

3. Secondary Outcome: Overall Survival
Description: Analyzed using the Kaplan-Meier method.
Time Frame: Up to 2 years
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Treatment (Tivantinib)
Number analyzed (Participants) | 18
Months | 12.2 [7.1 to 22.2]

4. Secondary Outcome: Progression-free Survival
Description: Time to disease progression or death from any cause. Analyzed using the Kaplan-Meier method.
Time Frame: Up to 2 years
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Treatment (Tivantinib)
Number analyzed (Participants) | 18
Months | 1.9 [1.8 to 5.4]

5. Other Pre Specified Outcome: Change in Baseline Levels of Continuous or Ordinal Markers (e.g., Serum HGF/MET IHC) Between Responders and Non-responders
Description: Fisher's exact test will be performed for binary variables (e.g., presence/absence of MET gene amplification). Paired t-tests or Wilcoxon signed-ranks test, whichever is appropriate, will be used to examine the changes with treatment in the laboratory correlates that are continuous and McNemar's test will be used for binary markers.
Time Frame: Baseline to 1 year
Reporting Status: Not Posted

6. Other Pre Specified Outcome: Change in Serum HGF or MET IHC and Tumor Size Change (Percent Reduction in Sum of Longest Diameters)
Description: Will be evaluated by Spearman's rank correlation coefficient.
Time Frame: Baseline to 1 year
Reporting Status: Not Posted

7. Other Pre Specified Outcome: Association Between Baseline HGF, MET Gene Amplification, MET IHC and PFS
Description: Will be evaluated using the Cox regression model.
Time Frame: Baseline to 1 year
Reporting Status: Not Posted

ADVERSE EVENTS:
Arm/Group | Treatment (Tivantinib)
Serious Adverse Events (participants affected / at risk) | 3/18
Other Adverse Events (participants affected / at risk) | 17/18
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Treatment (Tivantinib) (N=18)
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 1
Lung infection (Respiratory, thoracic and mediastinal disorders) | 1
Pleuritic pain (Respiratory, thoracic and mediastinal disorders) | 1
Small intestinal obstruction (Gastrointestinal disorders) | 1
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Treatment (Tivantinib) (N=18)
Abdominal distension (Gastrointestinal disorders) | 1
Abdominal pain (Gastrointestinal disorders) | 2
Alanine aminotransferase increased (Investigations) | 3
Alkaline phosphaase increased (Investigations) | 2
Anemia (Blood and lymphatic system disorders) | 9
Anorexia (Metabolism and nutrition disorders) | 3
Anxiety (Psychiatric disorders) | 2
Aspartate aminotransferase increase (Investigations) | 5
Back pain (Musculoskeletal and connective tissue disorders) | 1
Blurred vision (Eye disorders) | 1
Bruising (Injury, poisoning and procedural complications) | 1
Chest wall pain (Musculoskeletal and connective tissue disorders) | 2
Chronic kidney disease (Renal and urinary disorders) | 1
Constipation (Gastrointestinal disorders) | 2
Cough (Respiratory, thoracic and mediastinal disorders) | 3
Creatinine increased (Investigations) | 4
Dehydration (Metabolism and nutrition disorders) | 1
Diarrhea (Gastrointestinal disorders) | 4
Dizziness (Nervous system disorders) | 1
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 7
Ear pain (Ear and labyrinth disorders) | 1
Edema (Respiratory, thoracic and mediastinal disorders) | 1
Fatigue (General disorders) | 14
Fever (General disorders) | 3
Flu like symptoms (General disorders) | 1
Gastroesophageal reflux disease (Gastrointestinal disorders) | 1
Jitteriness (General disorders) | 1
Headache (Nervous system disorders) | 2
Hypercalcemia (Metabolism and nutrition disorders) | 1
Hyperglycemia (Metabolism and nutrition disorders) | 1
Hyperkalemia (Metabolism and nutrition disorders) | 4
Hypertension (Vascular disorders) | 1
Hypoalbuminemia (Metabolism and nutrition disorders) | 5
Hypocalcemia (Metabolism and nutrition disorders) | 1
Hypokalemia (Metabolism and nutrition disorders) | 1
Hyponatremia (Metabolism and nutrition disorders) | 3
Hypophosphatemia (Metabolism and nutrition disorders) | 3
Hypotension (Vascular disorders) | 1
Lymphocyte count decreased (Investigations) | 1
Memory impairment (Nervous system disorders) | 1
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 1
Nausea/vomiting (Gastrointestinal disorders) | 3
Neuropathy-sensory (Nervous system disorders) | 2
Non-cardiac chest pain (General disorders) | 1
Pain (General disorders) | 4
Palpitations (Cardiac disorders) | 1
Platelet count decreased (Investigations) | 1
Presyncope (Nervous system disorders) | 1
Productive cough (Respiratory, thoracic and mediastinal disorders) | 1
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 1
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 1
Sinus bradycardia (Cardiac disorders) | 3
Sore throat (Respiratory, thoracic and mediastinal disorders) | 2
Testicular pain (Reproductive system and breast disorders) | 1
Urinary tract infection (Infections and infestations) | 1
White blood cell decreased (Investigations) | 4

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of 60 days or less